CLINICAL TRIAL: NCT03103490
Title: 18F-FSPG PET/MRI or PET/CT Imaging of Cardiac Sarcoidosis or Inflammation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Stanford University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Andrei Iagaru, Associate Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-40376
Record Dates: First submitted 2017-03-10; First posted 2017-04-06 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Sarcoidosis; Myocardial Inflammation
Keywords: PET/MR
MeSH Terms: conditions — Myocarditis | interventions — 4-(3-fluoropropyl)glutamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-FSPG (Other): Patients receive 18F-FSPG for detection of Cardiac Sarcoidosis or Inflammation
  Interventions: Drug: 18F-FSPG

INTERVENTIONS:
Drug: 18F-FSPG — Patients receive 8mCi of 18F-FSPG and undergo PET/MRI imaging (or PET/CT for patients with metal implants) to determine the ability of 18F-FSPG to localize to cardiac sarcoidosis or myocardial inflammation.

SUMMARY:
The investigators will evaluate the detection of cardiac sarcoidosis or inflammation using 18F-FSPG PET/MRI (or PET/CT for participants with metal implants).

DETAILED DESCRIPTION:
PET/MRI scans will be performed with a whole-body PET/MR imaging system capable of simultaneous PET and MR imaging (SIGNA, GE Healthcare, Milwaukee, WI). Approximately 45-60 minutes after IV injection of 8 mCi of 18F-FSPG, PET emission scanning and MRI acquisition T1 weighted scanning will begin imaging both whole body and the heart.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old at the time of the scan
* Patient with known or suspected cardiac sarcoidosis.
* Patient is capable of complying with study procedures
* Patient can remain still for duration of imaging procedure

Exclusion Criteria:

* Patient is pregnant or nursing
* Metallic implants (contraindicated for MRI)
* History of renal insufficiency (only for MRI contrast administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 participants signed consent; 28 were allocated to the study arm.
Groups:
- 18F-FSPG: Patients receive 18F-FSPG for detection of Cardiac Sarcoidosis or Inflammation using PET/MRI (or PET/CT for patients with metal implants).
Period: Overall Study
Arm/Group | 18F-FSPG
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18F-FSPG
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 20
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 18F-FSPG Uptake on PET/MRI or PET/CT Fused Images Indicating Cardiac Involvement of Sarcoidosis
Description: Diffuse (widespread), focal (point) and focal-on-diffuse (combination of the two) patterns of 18F-FSPG uptake will be considered to be positive findings indicating cardiac involvement of sarcoidosis or inflammation
Time Frame: average approximately 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-FSPG
Number analyzed (Participants) | 28
Participants | 2

2. Secondary Outcome: Number of Participants With Evidence of Whole Body 18F-FSPG Uptake on PET/MRI or PET/CT Fused Images Indicating Extra-cardiac Sarcoidosis
Description: The whole-body PET/MRI images will be evaluated for findings of extra-cardiac sarcoidosis. Evidence of 18F-FSPG uptake within the whole body will indicate a positive finding for the presence of extra-cardiac sarcoidosis.
Time Frame: average approximately 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-FSPG
Number analyzed (Participants) | 28
Participants | 11

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | 18F-FSPG
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03103490/Prot_000.pdf